CLINICAL TRIAL: NCT00002812
Title: Treatment of Patients With Acute Lymphoblastic Leukemia With Unfavorable Features: A Phase III Group-wide Study
Brief Title: Combination Chemotherapy in Treating Children With Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1961; CCG-1961 (Other: Children's Cancer Group); CDR0000064953 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-11-24 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Doxorubicin; Idarubicin; Mercaptopurine; Methotrexate; pegaspargase; Prednisone; Thioguanine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A - Standard BFM of Standard Duration (RER) (Experimental): Induction chemotherapy Days 0 - 7. Prednisone 60 mg/m² PO 4 x day. Vincristine sulfate 1.5 mg/m² IV push weekly x 2 Days 0 and 7. Daunomycin (daunorubicin hydrochloride) 25 mg/m² IV push (over 15 min.) weekly x 2 Days 0 and 7. IT Cytosine Arabinoside (cytarabine, Ara-C) Day 0. Asparaginase 6000 IU/m² IM x 3 Days 3, 5, and 7. Day 7 Bone Marrow. Consolidation (Phase II) (5 weeks) Prednisone Taper, cyclophosphamide, cytosine arabinoside (Ara-C), mercaptopurine, vincristine sulfate, pegaspargase, IT Methotrexate and radiation therapy.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: idarubicin; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Arm B - Standard BFM with Double Delayed Intensification (RER) (Experimental): Induction chemotherapy Days 0 - 7. Prednisone 60 mg/m² PO 4 x day. Vincristine sulfate 1.5 mg/m² IV push weekly x 2 Days 0 and 7. Daunomycin (daunorubicin hydrochloride) 25 mg/m² IV push (over 15 min.) weekly x 2 Days 0 and 7. IT Cytosine Arabinoside (cytarabine, Ara-C) Day 0. Asparaginase 6000 IU/m² IM x 3 Days 3, 5, and 7. Day 7 Bone Marrow Consolidation (5 weeks) (Phase II) Prednisone Taper, cyclophosphamide, cytosine arabinoside (Ara-C), mercaptopurine, vincristine sulfate, pegaspargase, IT Methotrexate and radiation therapy.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: idarubicin; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Arm C - Augumented BFM of Standard Duration (RER) (Experimental): Induction chemotherapy Days 0 - 7. Prednisone 60 mg/m² PO 4 x day. Vincristine sulfate 1.5 mg/m² IV push weekly x 2 Days 0 and 7. Daunomycin (daunorubicin hydrochloride) 25 mg/m² IV push (over 15 min.) weekly x 2 Days 0 and 7. IT Cytosine Arabinoside (cytarabine, Ara-C) Day 0. Asparaginase 6000 IU/m² IM x 3 Days 3, 5, and 7. Day 7 Bone Marrow Consolidation (9 weeks) (Phase II) Prednisone Taper, cyclophosphamide, cytosine arabinoside (Ara-C), mercaptopurine, vincristine sulfate, pegaspargase, IT Methotrexate and radiation therapy.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: idarubicin; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy
- Arm D - Augmented BFM with Dbl Delayed Intensification (RER) (Experimental): Induction chemotherapy Days 0 - 7. Prednisone 60 mg/m² PO 4 x day. Vincristine sulfate 1.5 mg/m² IV push weekly x 2 Days 0 and 7. Daunomycin (daunorubicin hydrochloride) 25 mg/m² IV push (over 15 min.) weekly x 2 Days 0 and 7. IT Cytosine Arabinoside (cytarabine, Ara-C) Day 0. Asparaginase 6000 IU/m² IM x 3 Days 3, 5, and 7. Day 7 Bone Marrow Consolidation (9 weeks) (Phase II) Prednisone Taper, cyclophosphamide, cytosine arabinoside (Ara-C), mercaptopurine, vincristine sulfate, pegaspargase, IT Methotrexate and radiation therapy.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: idarubicin; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: asparaginase — Given IV
  Other Names: E. coli; Elspar; NSC-109229
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC-26271
Drug: cytarabine — Given IV
  Other Names: Cytosine Arabinoside; Ara-C; Cytosar-U; NSC-63878
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Daunomycin Hydrochloride; Cerrubidine; NSC-82151
Drug: dexamethasone — Given IV
  Other Names: Decadron; NSC-34521
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin; NSC-123127
Drug: idarubicin — Given IV
  Other Names: Idarubicin Hydrochloride; Idamycin; NSC-256439
Drug: mercaptopurine — Given IV
  Other Names: 6-MP; Purinethol; NSC-755
Drug: methotrexate — Given PO
  Other Names: NSC-740
Drug: pegaspargase — Given IV
  Other Names: Asparaginase; Oncaspar
Drug: prednisone — Given PO
  Other Names: NSC-10023
Drug: thioguanine — Given IV
  Other Names: 6-TG; NSC-752
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; NSC-67574
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug and giving the drugs in different combinations may kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of standard combination chemotherapy treatment with more intensive combination chemotherapy in treating children with acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the outcomes in children with higher risk acute lymphocytic leukemia (ALL) treated with postinduction chemotherapy based on marrow response on day 7 of induction therapy: for patients with rapid early response (M1/M2), standard vs intensified consolidation chemotherapy and standard vs prolonged duration of intensification chemotherapy; for patients with slow early response, addition of doxorubicin vs idarubicin and cyclophosphamide to intensification chemotherapy. II. Decrease the incidence of avascular necrosis by alternating dexamethasone dosing in patients undergoing 2 courses of delayed intensification. III. Assess the impact of day 7 marrow status on outcome in these patients. IV. Determine prognosis more precisely by supplementing presenting clinical features, immunophenotype, ploidy, cytogenetics, and early marrow response with BAX/BCL-2 ratios, pattern of tyrosine kinase activation, leukemic burden following induction and intensification therapy, and development of high antibody titer to E. coli asparaginase. V. Correlate the traditional prognostic factors of day 7 marrow response, immunophenotype, ploidy, cytogenetics, and early marrow response with BAX/BCL-2 ratios.

OUTLINE: This is a partially randomized, multicenter study. Patients are stratified by center. Patients receive one course of the VPLD regimen comprised of vincristine IV and daunorubicin IV over 15 minutes to 2 hours on days 0 and 7, oral prednisone daily on days 0-7, intrathecal cytarabine on day 0, and asparaginase or pegaspargase intramuscularly on days 3, 5, and 7. Patients are assigned to 1 of 2 two postinduction chemotherapy groups based on bone marrow response on day 7 of induction. Patients with M1/M2 marrow on day 7 are considered rapid early responders. Patients with M3 marrow on day 7 are considered slow early responders. Group 1: Rapid early responders Patients receive 2 additional courses of VPLD induction chemotherapy. Patients are then randomized to 1 of 4 treatment arms: Arm I: Beginning on day 35 of induction therapy, patients receive standard Berlin-Frankfurt-Munster (BFM) regimen with standard delayed intensification. Standard BFM for patients in arm I consists of the following: consolidation over 5 weeks with cyclophosphamide, cytarabine, and mercaptopurine; interim maintenance over 8 weeks with oral methotrexate and mercaptopurine (MTX/MP); and delayed intensification over 7 weeks consisting of reinduction with vincristine, doxorubicin, oral dexamethasone, and asparaginase or pegaspargase followed by reconsolidation with cyclophosphamide, thioguanine, and cytarabine. Arm II: Patients receive standard BFM regimen with double delayed intensification. Patients receive therapy similar to those in arm I, but dexamethasone is interrupted for 1 week during delayed intensification and the intensification regimen is repeated, separated by an 8 week interim maintenance course of oral MTX/MP. Arm III: Patients receive augmented BFM regimen with standard delayed intensification. Patients receive 9 weeks of consolidation therapy with 2 courses of vincristine and pegaspargase alternating with the arm I consolidation therapy. Vincristine, intravenous methotrexate, and pegaspargase (the Capizzi I regimen) are substituted for oral MTX/MP in the interim maintenance regimen. Pegaspargase is substituted for asparaginase and two additional doses of vincristine are administered during delayed intensification. Arm IV: Patients receive augmented BFM regimen with double delayed intensification. Patients receive intensified chemotherapy throughout, combining the additional therapy given to patients in arms II and III. Patients receiving augmented BFM regimen receive pegaspargase instead of asparaginase. Patients with CNS disease at diagnosis are treated only on arm IV. Patients who are Philadelphia chromosome positive and do not have a bone marrow donor are nonrandomly assigned to the treatment group for slow early responders. All RER patients receive the same maintenance therapy with vincristine/prednisone and oral MTX/MP. Intrathecal methotrexate is administered periodically throughout protocol treatment. Group 2: Slow early responders Patients receive augmented BFM consolidation therapy and Capizzi I interim maintenance identical to that received by rapid early responders in arm IV. Patients are then randomized to receive double delayed intensification with either idarubicin or doxorubicin and concurrent cyclophosphamide. All patients receive the same maintenance therapy with vincristine/prednisone and oral MTX/MP. Intrathecal MTX is administered periodically throughout protocol treatment. Patients with CNS disease at entry receive craniospinal irradiation daily for 5 consecutive days beginning on day 0 of consolidation therapy. All slow early responders at diagnosis receive cranial irradiation daily for 5 consecutive days during consolidation therapy. Patients with testicular leukemia at diagnosis receive bilateral testicular irradiation daily for 5 consecutive days during consolidation chemotherapy. Groups 1 and 2: Maintenance therapy continues for 2 years for girls or 3 years for boys beyond completion of consolidation therapy. Patients are followed every 4-6 weeks for 1 year, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 1,520 patients will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute lymphocytic leukemia (ALL) with M3 bone marrow No FAB L3 morphology CNS or overt testicular leukemia at diagnosis allowed High risk status 10-21 years old with any white blood count (WBC) 1-9 years old with WBC of 50,000/mm3 or greater

PATIENT CHARACTERISTICS: Age: 1 to 21 Performance status: Not specified Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: No prior therapy for ALL except: Emergency therapy for blast crisis, superior vena cava syndrome, or renal failure due to leukemic infiltration Biologic therapy: Not specified Chemotherapy: Intrathecal cytarabine or methotrexate allowed at diagnostic lumbar puncture Induction therapy must begin within 72 hours after intrathecal injection Endocrine therapy: At least 1-2 months since prior prednisone, for less than 48 hours, for reactive airway disease Inhalational steroids allowed Radiotherapy: Not specified Surgery: Not specified

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2078 (Actual)
Dates: Start 1996-09; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | from the time of randomization where the life table events will consist of the first occurrence of the following events: failure to achieve remission, leukemic relapse at any site, death, or occurrence of a second malignancy.
  The primary outcome index used in examining most of the randomized treatment groups will be event-free survival (EFS).

CONTACTS AND LOCATIONS:
Overall Officials: Nita L. Seibel, MD, Study Chair — Children's National Research Institute
Locations (35):
- United States (32):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Background] Nguyen K, Devidas M, Cheng SC, La M, Raetz EA, Carroll WL, Winick NJ, Hunger SP, Gaynon PS, Loh ML; Children's Oncology Group. Factors influencing survival after relapse from acute lymphoblastic leukemia: a Children's Oncology Group study. Leukemia. 2008 Dec;22(12):2142-50. doi: 10.1038/leu.2008.251. Epub 2008 Sep 25. PMID 18818707
- [Background] Butturini AM, Dorey FJ, Lange BJ, Henry DW, Gaynon PS, Fu C, Franklin J, Siegel SE, Seibel NL, Rogers PC, Sather H, Trigg M, Bleyer WA, Carroll WL. Obesity and outcome in pediatric acute lymphoblastic leukemia. J Clin Oncol. 2007 May 20;25(15):2063-9. doi: 10.1200/JCO.2006.07.7792. PMID 17513811
- [Background] Avramis VI, Panosyan EH. Pharmacokinetic/pharmacodynamic relationships of asparaginase formulations: the past, the present and recommendations for the future. Clin Pharmacokinet. 2005;44(4):367-93. doi: 10.2165/00003088-200544040-00003. PMID 15828851
- [Background] Seibel NL, Asselin BL, Nachman JB, et al.: Treatment of high risk T-cell acute lymphoblastic leukemia (T-ALL): comparison of recent experience of the Children's Cancer Group (CCG) and Pediatric Oncology Group (POG). [Abstract] Blood 104 (11): A-681, 2004.
- [Result] Arce FJ, Seibel N, Gaynon PS, et al.: Pharmacokinetics and pharmacodynamics of asparaginases in antibody-negative pediatric patients with higher risk acute lymphoblastic leukemia (ALL): a report from CCG-1961. [Abstract] J Clin Oncol 24 (Suppl 18): A-9027, 508s, 2006.
- [Result] Avramis VI, Ettinger L, Martin-Aragon S, et al.: Anti-asparaginase (ASNase) antibody (Ab) in pediatric patients in high risk ALL study (CCG-1961): correlation of Ab and clinical allergy. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A2319, 2000.
- [Result] Avramis VI, Panosyan E, Avramis IA, et al.: Anti-asparaginase (ASNase) antibody (Ab) and ASNase activity in children with higher risk acute lymphoblastic leukemia (HR ALL) (CCG-1961). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1592, 2002.
- [Result] Bhojwani D, Kang H, Menezes RX, Yang W, Sather H, Moskowitz NP, Min DJ, Potter JW, Harvey R, Hunger SP, Seibel N, Raetz EA, Pieters R, Horstmann MA, Relling MV, den Boer ML, Willman CL, Carroll WL; Children's Oncology Group Study; Dutch Childhood Oncology Group; German Cooperative Study Group for Childhood Acute Lymphoblastic Leukemia. Gene expression signatures predictive of early response and outcome in high-risk childhood acute lymphoblastic leukemia: A Children's Oncology Group Study [corrected]. J Clin Oncol. 2008 Sep 20;26(27):4376-84. doi: 10.1200/JCO.2007.14.4519. PMID 18802149
- [Result] Dhall G, Jones T, Radvinsky D, et al.: Adverse reactions to PEG and Erwinia asparaginase and correlation with anti-asparaginase antibody data and survival in children with acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group study CCG 1961. [Abstract] Blood 114 (22): A-3077, 2009.
- [Result] Dhall G, Robison NJ, Rubin JI, et al.: Incidence of adverse reactions to post-induction asparaginase (ASP) therapy in children and adolescents with high-risk acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group Study CCG-1961. [Abstract] J Clin Oncol 26 (Suppl 15): A-10021, 2008.
- [Result] Freyer DR, Devidas M, La M, Carroll WL, Gaynon PS, Hunger SP, Seibel NL. Postrelapse survival in childhood acute lymphoblastic leukemia is independent of initial treatment intensity: a report from the Children's Oncology Group. Blood. 2011 Mar 17;117(11):3010-5. doi: 10.1182/blood-2010-07-294678. Epub 2010 Dec 30. PMID 21193696
- [Result] Freyer DR, Seibel NL, La MK, et al.: Survival after relapse in higher risk acute lymphoblastic leukemia (ALL) in children and adolescents is independent of prior treatment intensity: a report from the Children's Oncology Group (COG). [Abstract] Blood 112 (11): A-917, 2008.
- [Result] Hastings C, Sather HN, Seibel NL, et al.: Outcomes in children and adolescents with a markedly elevated white blood cell count (>200,000) at diagnosis of high risk acute lymphoblastic leukemia (ALL): a report from the Children's Oncology Group. [Abstract] Blood 108 (11): A-1870, 2006.
- [Result] Hastings C, Whitlock JA, La M, et al.: Improved outcome of children with Down syndrome (DS) and high risk acute lymphocytic leukemia (HR-ALL): a report of CCG-1961. [Abstract] Blood 110 (11): A-586, 2007.
- [Result] Henze G. Early postinduction intensification therapy is essential in childhood acute lymphoblastic leukemia. Nat Clin Pract Oncol. 2008 Sep;5(9):502-3. doi: 10.1038/ncponc1184. Epub 2008 Jul 22. PMID 18648353
- [Result] Mattano LA Jr, Devidas M, Nachman JB, Sather HN, Hunger SP, Steinherz PG, Gaynon PS, Seibel NL; Children's Oncology Group. Effect of alternate-week versus continuous dexamethasone scheduling on the risk of osteonecrosis in paediatric patients with acute lymphoblastic leukaemia: results from the CCG-1961 randomised cohort trial. Lancet Oncol. 2012 Sep;13(9):906-15. doi: 10.1016/S1470-2045(12)70274-7. Epub 2012 Aug 15. PMID 22901620
- [Result] Nachman JB, La MK, Hunger SP, Heerema NA, Gaynon PS, Hastings C, Mattano LA Jr, Sather H, Devidas M, Freyer DR, Steinherz PG, Seibel NL. Young adults with acute lymphoblastic leukemia have an excellent outcome with chemotherapy alone and benefit from intensive postinduction treatment: a report from the children's oncology group. J Clin Oncol. 2009 Nov 1;27(31):5189-94. doi: 10.1200/JCO.2008.20.8959. Epub 2009 Oct 5. PMID 19805689
- [Result] Nachman J, Siebel N, Sather H, et al.: Outcome for adolescent and young adults 16-21 years of age (AYA) with acute lymphoblastic leukemia (ALL) treated on the Children' s Cancer Group (CCG) 1961 study. [Abstract] Blood 104 (11): A-683, 2004.
- [Result] Panosyan EH, Grigoryan RS, Avramis IA, Seibel NL, Gaynon PS, Siegel SE, Fingert HJ, Avramis VI. Deamination of glutamine is a prerequisite for optimal asparagine deamination by asparaginases in vivo (CCG-1961). Anticancer Res. 2004 Mar-Apr;24(2C):1121-5. PMID 15154634
- [Result] Panosyan EH, Seibel NL, Grigoryan RS, et al.: Pharmacokinetics and pharmacodynamics of three asparaginases in pediatric patients with higher risk acute lymphoblastic leukemia: a report from CCG-1961. [Abstract] Blood 104 (11): A-2745, 2004.
- [Result] Panosyan EH, Seibel NL, Martin-Aragon S, Gaynon PS, Avramis IA, Sather H, Franklin J, Nachman J, Ettinger LJ, La M, Steinherz P, Cohen LJ, Siegel SE, Avramis VI; Children's Cancer Group Study CCG-1961. Asparaginase antibody and asparaginase activity in children with higher-risk acute lymphoblastic leukemia: Children's Cancer Group Study CCG-1961. J Pediatr Hematol Oncol. 2004 Apr;26(4):217-26. doi: 10.1097/00043426-200404000-00002. PMID 15087948
- [Result] Seibel NL, Steinherz PG, Sather HN, Nachman JB, Delaat C, Ettinger LJ, Freyer DR, Mattano LA Jr, Hastings CA, Rubin CM, Bertolone K, Franklin JL, Heerema NA, Mitchell TL, Pyesmany AF, La MK, Edens C, Gaynon PS. Early postinduction intensification therapy improves survival for children and adolescents with high-risk acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood. 2008 Mar 1;111(5):2548-55. doi: 10.1182/blood-2007-02-070342. Epub 2007 Nov 26. PMID 18039957
- [Result] Withycombe JS, Post-White JE, Meza JL, Hawks RG, Smith LM, Sacks N, Seibel NL. Weight patterns in children with higher risk ALL: A report from the Children's Oncology Group (COG) for CCG 1961. Pediatr Blood Cancer. 2009 Dec 15;53(7):1249-54. doi: 10.1002/pbc.22237. PMID 19688832